CLINICAL TRIAL: NCT04674800
Title: A Multi Center, Extension Study to Evaluate the Safety and Efficacy of MYL-1701P in Subjects With Diabetic Macular Edema Completed MYL-1701P-3001 Study.
Brief Title: Extension Study of MYL-1701P-3001 for Safety and Efficacy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Collaborators: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFIL-IJZ-3002
Record Dates: First submitted 2020-11-30; First posted 2020-12-19 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; BCVA; ETDRS Letters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single, test arm (Experimental): MYL-1701P- Subjects will receive 3 doses each of 2 mg at 8 weeks interval
  Interventions: Biological: MYL-1701P, a proposed biosimilar to Eylea

INTERVENTIONS:
Biological: MYL-1701P, a proposed biosimilar to Eylea — Open label and single arm

SUMMARY:
This Study (AFIL-IJZ-3002) is designed to evaluate the safety, efficacy and immunogenicity of MYL-1701P among a group of participants successfully completing MYL-1701P-3001 study.

DETAILED DESCRIPTION:
Diabetic retinopathy is an important cause of blindness worldwide. The International Diabetes Federation estimates that 285 million people worldwide have diabetes mellitus and approximately 7% of these individuals are affected by diabetic macular edema.

EYLEA® (aflibercept) injection, an anti-Vascular Endothelial Growth Factor (VEGF) agent, has been approved by the FDA and EMA for the treatment of Diabetic Macular Edema (DME).

Mylan Inc. and Momenta Pharmaceuticals, Inc. are developing MYL-1701P, a proposed biosimilar to Eylea.

MYL-1701P-3001 study was designed to evaluate the efficacy, safety, pharmacokinetics, and immunogenicity of MYL-1701P in the treatment of subjects with Diabetic Macular Edema (DME). Eligible subjects from MYL-1701P-3001 study will be enrolled in the AFIL-IJZ-3002 study. All enrolled subjects will receive three doses of MYL-1701P every eight weeks. Subjects will attend the clinic visits for safety and efficacy assessments including BCVA, SD-OCT, complete ophthalmological examinations during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject participated in the MYL-1701P-3001 study
2. Subject requires treatment with intravitreal anti-VEGF therapy
3. Subject is able to understand and voluntarily provide written informed consent to participate in the study.
4. If female of childbearing potential, the subject must have negative pregnancy tests and should not be nursing or planning a pregnancy.
5. Subject is willing to comply with the study duration, study visits and study related procedures.
6. If female, subject must be:

   * Surgically sterilized via hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; or
   * Of childbearing potential and practicing an acceptable form of birth control
   * Of non-childbearing potential
7. If male, subject must be surgically or biologically sterile. If not sterile, the subject must agree to use an acceptable form of birth control

Exclusion Criteria:

1. Subjects with known hypersensitivity to aflibercept or any of the excipients
2. Subjects will be excluded if any of the following conditions are met in the study eye:

   * Subjects with active ocular inflammation.
   * Subjects with uncontrolled glaucoma
   * Surgery for glaucoma in the past or likely to be needed in the future.
3. Subjects with active or suspected ocular or periocular infection including but not limited to infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye.
4. Subjects who plan to participate in another clinical study while enrolled in this study.
5. Subjects receiving treatment for a serious systemic infection.
6. Subjects with uncontrolled hypertension defined as systolic blood pressure > 160 mm Hg or diastolic blood pressure > 95 mm Hg.
7. Subjects with a history of cerebrovascular accident or myocardial infarction within 6 months of enrollment.
8. Subjects with renal failure requiring dialysis or renal transplant.
9. Subjects with a history or presence of any clinically significant condition, that in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment emergent adverse events (TEAEs). | Week 20
  Number of participants with TEAEs

SECONDARY OUTCOMES:
Change from baseline in BCVA | Weeks 8, 16 and 20
  Best Corrected Visual Acuity (BCVA) will be assessed by Early Treatment Diabetic Retinopathy Letters (ETDRS)
Change from baseline in CRT | Weeks 8, 16 and 20
  Central retinal thickness (CRT) will be evaluated using spectral-domain-optical coherence tomography (SD-OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Prasanna Ganapathi, MD, Study Director — Mylan Inc.
Locations (15):
- India (15):
  - Mylan Investigative site, Hyderabad, Andhra Pradesh
  - Mylan Investigative Site, Visakhapatnam, Andhra Pradesh
  - Mylan Investigative Site, Ahmedabad, Gujarat
  - Mylan Investigative site, Ahmedabad, Gujarat
  - Mylan Investigative site, Bangalore, Karnataka
  - Mylan Investigative Site, Bangalore, Karnataka
  - Mylan Investigative Site, Bengaluru, Karnataka
  - Mylan Investigative Site, Mumbai, Maharashtra
  - Mylan Investigative site, Bhubaneswar, Odisha
  - Mylan Investigative Site, Chandigarh, Punjab
  - Mylan Investigative site, Jaipur, Rajasthan
  - Mylan Investigative site, Madurai, Tamil Nadu
  - Mylan Investigative site, Tirunelveli, Tamil Nadu
  - Mylan Investigative Site, Noida, Uttar Pradesh
  - Mylan Investigative site, New Delhi

IPD SHARING:
Plan to Share IPD: No